CLINICAL TRIAL: NCT02232815
Title: A Randomized Multicentre Trial to Compare Outcomes for Patients With Ischaemic Heart Disease and Bifurcation Coronary Artery Lesions Who Are Treated With Xience or Synergy Stents
Brief Title: CELTIC Bifurcation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Cardiovascular Research Center (Network)
Collaborators: Ceric Sàrl (Industry)
Responsible Party: Sponsor
Other Study IDs: BSC-02
Record Dates: First submitted 2014-08-25; First posted 2014-09-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Bifurcations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine outcomes for patients treated by planned culotte stenting and compare outcomes with 2 different stent platforms, the next generation Synergy II and the Xience Xpedition DES platforms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient >18 years old
* Females of childbearing potential with a negative pregnancy test
* Coronary artery disease requiring revascularization that is amenable to PCI
* Medina 1,1,1 bifurcation lesion [13] with >70% lesion in both the main vessel and the side branch by visual assessment
* Main branch and side branch ≥ 2.5mm in diameter by visual assessment
* Both vessels require stenting in the opinion of the operator

Exclusion Criteria:

* Acute myocardial infarction with ongoing ST-elevation
* Cardiogenic shock
* Lesion involves the left main coronary artery
* Lesion involves bypass graft
* Plan to treat >1 other coronary vessel at the time of inclusion
* Chronic total occlusion of any target vessel
* Left ventricular ejection fraction <20%
* Requirement for ongoing haemodialysis
* Life-expectancy limited to <12 months due to co-morbid condition
* Known allergy to Aspirin
* Known allergy to Clopidorel and Prasugrel and Ticagrelor
* Known allergy to stent drug elutant
* Known allergy to any other component of either the Synergy II or Xience Xpedition stents systems
* Ongoing participation in another investigational device or drug study
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planed for culotte DES stenting
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite measure of Adverse events | 9 months
  Composite of:
  * Death
  * Myocardial Infarction
  * CVA
  * Target Vessel Failure (Composite of Target Vessel Revascularization and Target Vessel Inadequacy)
  * Definite or Probable stent thrombosis (ARC criteria [14])
  * Binary angiographic restenosis

SECONDARY OUTCOMES:
Technical success (deployment of stents in both branches with <20% residual stenosis and kissing balloon inflation at end of procedure) | Day 0, during procedure
Total procedure time | Day 0, during procedure
Total radiation dose | Day 0, during procedure
Need to use secondary equipment or manoeuvres to complete the case | Day 0, during procedure
  extra support guidewires, anchor balloons or mother & daughter catheter
Evidence of longitudinal stent compression at index implantation | Day 0, during procedure
Evidence of stent fracture at angiographic follow-up | Day 0, during procedure
Composite measure of Adverse events | 24 months
  Composite of:
  * Death
  * Myocardial Infarction
  * CVA
  * Target Vessel Failure (Composite of Target Vessel Revascularization and Target Vessel Inadequacy)
  * Definite or Probable stent thrombosis (ARC criteria [14])

CONTACTS AND LOCATIONS:
Locations (6):
- St Vincent's Hospital Dublin, Dublin, Ireland
- United Kingdom (5):
  - Belfast Health & Social Care Trust, Belfast
  - Bristol Royal Inﬁrmary, Bristol
  - Edinburgh Royal Inﬁrmary, Edinburgh
  - Golden Jubilee, Glasgow
  - Kings College, London